CLINICAL TRIAL: NCT01504711
Title: Prevention of Nausea and Vomiting Secondary to FOLFIRINOX Chemotherapy in Gastrointestinal Cancer Patients
Brief Title: Fosaprepitant Dimeglumine in Preventing Nausea and Vomiting in Patients With Gastrointestinal Cancer Receiving Combination Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Philip (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Philip Philip, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-116; NCI-2011-03735 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30 CA022453I (Other: National Institutes of Health); P30CA022453 (NIH)
Record Dates: First submitted 2011-12-22; First posted 2012-01-05 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-09

CONDITIONS: Gastrointestinal Cancer; Nausea Post Chemotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — fosaprepitant; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nausea and vomiting prophylaxis) (Experimental): Receive fosaprepitant dimeglumine IV 30 mins. prior to FOLFIRINOX chemotherapy.
  Interventions: Drug: fosaprepitant dimeglumine

INTERVENTIONS:
Drug: fosaprepitant dimeglumine — Given IV
  Other Names: EMEND®

SUMMARY:
This clinical trial studies fosaprepitant dimeglumine in preventing nausea and vomiting in patients with gastrointestinal cancer receiving combination chemotherapy. Antiemetic drugs, such as fosaprepitant dimeglumine, may help lessen or prevent nausea and vomiting in patients treated with chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate efficacy of the addition of fosaprepitant (fosaprepitant dimeglumine) in controlling acute and delayed vomiting with the standard prophylactic anti-emetic combination of 5-HT3 receptor antagonist and dexamethasone for gastrointestinal cancer patients receiving FOLFIRINOX (5-FU [fluorouracil], oxaliplatin and irinotecan [irinotecan hydrochloride]) chemotherapy.

II. To determine the rate of complete response (no emetic episode and no rescue medication) in the combined acute and delayed phase from 0-120 hours after chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the incidence of nausea and vomiting in both acute (< 24 hours) and delayed (24- 120 hours) setting in patients receiving FOLFIRINOX chemotherapy.

TERTIARY OBJECTIVES:

I. Follow overall survival in patients receiving FOLFIRINOX chemotherapy.

OUTLINE:

Patients receive fosaprepitant dimeglumine intravenously (IV) 30 minutes prior to FOLFIRINOX chemotherapy.

After completion of study treatment, patients are followed up for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving FOLFIRINOX chemotherapy
* Southwest Oncology Group (SWOG) Performance status 0 or 1
* Ability of patient or guardian to understand and to provide voluntary written informed consent

Exclusion Criteria:

* Patient with current illness requiring chronic systemic steroids use or requiring chronic use of anti emetics
* Patients with gastrointestinal (GI) obstruction or active peptic ulcer disease who cannot take oral medication
* Known hypersensitivity to any component of the study regimen
* Patients taking any of the following medications: Oral contraceptives (except for the administration of stopping menses), tolbutamide, phenytoin, midazolam, ketoconazole, rifampin, paroxetine, and Diltiazem
* Pregnant or nursing women
* Patients using illegal drugs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2016-12-29 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, M.D., Ph.D., F.R.C.P, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nausea and Vomiting Prophylaxis)
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 30 patients were eligible and consented to this protocol. 3 of these patients never began treatment, leaving our final analysis number at 27.
Arm/Group | Treatment (Nausea and Vomiting Prophylaxis)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Control of Vomiting and Rescue Medication Control
Description: Achieved if a patient has no episodes of vomiting and requires no rescue medication during the first 120 hours after fosaprepitant dimeglumine administration.
Time Frame: From 0-120 hours after first course of chemotherapy
Population: The analysis set includes patients (n=26) who returned an outcomes diary at 24 or 120 hours post treatment. 1 patient could not be evaluated as they did not return their diary.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nausea and Vomiting Prophylaxis)
Number analyzed (Participants) | 26
percentage of participants | 26.9 [15.3 to 42.9]

2. Secondary Outcome: Percentage of Participants With Control of Both Acute and Delayed Vomiting
Description: Achieved if a patient has no episodes of vomiting at both 24 and 120 hours after fosaprepitant dimeglumine administration.
Time Frame: in approximately 28 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nausea and Vomiting Prophylaxis)
Number analyzed (Participants) | 26
percentage of participants | 65.4 [49.3 to 78.6]

3. Secondary Outcome: Percentage of Participants With Control of Both Acute and Delayed Nausea
Description: Achieved if a patient has no episodes of nausea at both 24 and 120 hours after fosaprepitant dimeglumine administration.
Time Frame: in approximately 28 months
Population: The analysis set includes patients (n=25) who returned an outcomes diary at 24 or 120 hours post treatment with nausea information filled out. 2 patients could not be evaluated as they did not return their diary with nausea information filled out.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nausea and Vomiting Prophylaxis)
Number analyzed (Participants) | 25
percentage of participants | 28.0 [16.0 to 44.3]

4. Secondary Outcome: Overall Survival
Time Frame: Time of initiation of treatment until death or censor assessed up to 26 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nausea and Vomiting Prophylaxis)
Number analyzed (Participants) | 27
months | 11.5 [4.8 to 15.5]

ADVERSE EVENTS:
Time Frame: The adverse event information includes unexpected and/or serious adverse events from cycles 1 and 2 of treatment. As each cycle last approximately 2 weeks, the adverse event information in this report covers the first month of treatment. The mortality information includes death events while the patients were on treatment or in follow-up (up to 27 months).
Groups:
- All Participants: All participants
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 22/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=27)
GI bleed from gastric ulcer (Gastrointestinal disorders) | 1
Uncontrolled nausea (Gastrointestinal disorders) | 1
bowel obstruction (Gastrointestinal disorders) | 1
intractable nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=27)
Vomiting (Gastrointestinal disorders) | 4
Hypokalemia (General disorders) | 3
Dehydration (General disorders) | 3
Anemia (General disorders) | 3
Hyponatremia (General disorders) | 2
Decreased white blood cell count (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT01504711/Prot_SAP_000.pdf